CLINICAL TRIAL: NCT07315035
Title: A Randomized, Controlled, Phase-II Trial of Neoadjuvant QL1706 (Iparomlimab /Tuvonralimab) Combined With SOX Versus SOX Alone Followed by Curative Gastrectomy in Patients With Locally Advanced Diffuse-Type Gastric Adenocarcinoma
Brief Title: QL1706-SOX vs SOX Alone as Neoadjuvant Therapy for Resectable Diffuse-Type Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Affiliated Jiangning Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QILIN-01
Record Dates: First submitted 2025-12-05; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer Stage III
Keywords: QL1706; Diffused-type Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-center, parallel-group, superiority trial with a two-arm randomized design. After confirmation of eligibility, participants are allocated 1:1 by central computer-generated randomization (block size 4, stratified by baseline ECOG performance status 0 vs 1) to receive either QL1706 plus SOX (experimental arm) or SOX alone (control arm) as neoadjuvant therapy. Randomization is open-label; however, pathological response and surgical margin status are assessed by two independent gastrointestinal pathologists blinded to treatment assignment. No crossover is permitted. The study schema is fixed: three to four 3-week cycles of protocol-specified therapy, mandatory restaging within 2 weeks after cycle 3, and curative-intent gastrectomy scheduled 4-6 weeks after the last dose. Post-operative adjuvant therapy is investigator-determined and recorded, but does not influence the primary endpoint analysis. This model allows direct comparison of immune-chemotherapy versus chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706+SOX (Experimental): QL1706 (Iparomlimab/Tuvonralimab) 5 mg/kg intravenous infusion on day 1 plus SOX (S-1 40-60 mg orally twice daily days 1-14 and oxaliplatin 130 mg/m² intravenous infusion on day 1) every 3 weeks for 3-4 cycles before curative gastrectomy.
  Interventions: Drug: QL1706 (Iparomlimab/Tuvonralimab); Drug: SOX Chemotherapy
- SOX (Active Comparator): S-1 40-60 mg orally twice daily days 1-14 and oxaliplatin 130 mg/m² intravenous infusion on day 1 every 3 weeks for 3-4 cycles before curative-intent gastrectomy.
  Interventions: Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: QL1706 (Iparomlimab/Tuvonralimab) — QL1706 is a first-in-class, fixed-ratio bispecific monoclonal antibody produced in a single Chinese hamster ovary cell line that simultaneously targets PD-1 (IgG4 framework) and CTLA-4 (IgG1 framework) with an approximate 2:1 molar ratio. This molecular design delivers dual immune checkpoint blockade in one infusion, distinguishing it from separate-agent combinations such as nivolumab plus ipilimumab. In this study QL1706 is given at 5 mg/kg (actual body weight) as a 60-minute intravenous infusion on day 1 of each 21-day cycle, immediately followed by oxaliplatin 130 mg/m² (2-hour infusion) and oral S-1 (40-60 mg bid days 1-14). The sequence is repeated for 3-4 cycles before planned surgery; no intra-patient dose escalation or reduction is allowed, but infusion may be delayed ≤12 weeks for immune-related adverse events. The comparator arm receives identical SOX chemotherapy without any investigational antibody, ensuring that any difference in pathological outcome can be attributed spec
  Arms: QL1706+SOX
Drug: SOX Chemotherapy — SOX chemotherapy consists of oxaliplatin 130 mg/m² delivered as a 2-hour intravenous infusion on day 1 plus oral S-1 (tegafur 40-60 mg, gimeracil and oteracil potassium in fixed 1:0.4:1 molar ratio) taken twice daily on days 1-14 of a 21-day cycle, repeated for 3-4 cycles before curative-intent gastrectomy. The S-1 dose is calculated by body-surface area: <1.25 m² → 40 mg, 1.25-1.5 m² → 50 mg, >1.5 m² → 60 mg per administration.

SUMMARY:
The goal of this randomized, open-label, phase II clinical trial is to determine whether adding the PD-1/CTLA-4 bispecific antibody QL1706 to standard SOX chemotherapy increases the pathological complete response rate in adults aged 18-75 years with resectable, locally advanced, diffuse-type, HER2-negative gastric adenocarcinoma (cT3-4aNxM0). Participants will be randomly assigned (1:1) to receive 3-4 neoadjuvant cycles of QL1706 plus SOX or SOX alone every 3 weeks, followed by curative-intent gastrectomy with D2 lymphadenectomy, and will be monitored post-operatively every 3 months for 2 years and every 6 months thereafter for recurrence, survival, and safety.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diffuse-type gastric adenocarcinoma (Lauren classification) with signet-ring cells ≥ 50 % of tumor volume HER2-negative by IHC or ISH per ASCO/CAP guidelines Clinical stage cT3-4aNxM0 (AJCC 8th ed.) on baseline EUS + contrast-enhanced CT/MRI; disease judged resectable by multidisciplinary team No prior gastric surgery, chemotherapy, radiotherapy, or immunotherapy for cancer Age 18-75 years; ECOG performance status 0-1 Adequate organ function (ANC ≥ 1.5 × 10⁹/L, platelet ≥ 100 × 10⁹/L, Hb ≥ 9 g/dL, ALT/AST ≤ 2.5 × ULN, TBIL ≤ 1.5 × ULN, creatinine ≤ 1.5 × ULN and calculated CrCl ≥ 60 mL/min, INR/PT ≤ 1.5 × ULN) within 14 days before randomization Left-ventricular ejection fraction ≥ 50 % by echocardiography; no clinically significant ECG abnormalities Negative serum β-hCG pregnancy test ≤ 7 days of first dose for women of child-bearing potential; agreement to use effective contraception through 6 months post-surgery Life expectancy ≥ 6 months Signed informed consent; able to comply with study procedures and follow-up

Exclusion Criteria:

Mixed or intestinal Lauren histology; mucinous or hepatoid variants Active gastrointestinal bleeding or endoscopic evidence of major vessel invasion Other malignancy within 5 years (except curatively treated basal-cell carcinoma, cervical carcinoma in situ, or superficial bladder cancer) Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4, or other T-cell co-stimulatory/antagonist agents Autoimmune disease requiring systemic immunosuppression within 2 years (e.g., prednisone > 10 mg/day equivalent) Receipt of live vaccine ≤ 30 days before first dose Known HIV-positive, active hepatitis B (HBsAg+ and HBV-DNA > 200 IU/mL), or hepatitis C infection (HCV RNA positive) Active tuberculosis or history of incompletely treated TB Severe cardiovascular disease: NYHA class ≥ II heart failure, unstable angina, myocardial infarction ≤ 6 months, uncontrolled arrhythmia, or uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100 mmHg) Peripheral neuropathy ≥ grade 2 per NCI-CTCAE v5.0 Pulmonary disease requiring systemic steroids (e.g., ≥ grade 2 pneumonitis) or oxygen therapy Active infection requiring systemic antibiotics, antivirals, or antifungals ≤ 7 days before first dose Known hypersensitivity to oxaliplatin, fluoropyrimidines, or Chinese hamster ovary cell-derived products Pregnancy or lactation Concurrent participation in another interventional clinical trial Any condition that, in the investigator's opinion, would compromise safe completion of protocol therapy or accurate assessment of outcomes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Perioperative
  Pathological complete response (pCR) rate, defined as the proportion of participants who achieve ypT0N0 (absence of viable tumor cells in the resected primary tumor and all examined lymph nodes, Mandard TRG 1 or Becker grade 1) after completion of 3-4 cycles of protocol-specified neoadjuvant therapy and subsequent curative-intent gastrectomy, assessed by central review of H&E-stained slides according to AJCC 8th edition criteria within 4 weeks of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China